CLINICAL TRIAL: NCT01169870
Title: A Randomized Phase II Trial of Genexol-PM vs Paclitaxel in Anthracycline-pretreated Metastatic Breast Cancer Patients
Brief Title: Genexol-PM Versus Paclitaxel in Anthracycline-pretreated Metastatic Breast Cancer Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: withdrawn studies
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Jungsil Ro, Chief, Center for Clinical Trials, National Cancer Center, Korea, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-07-278
Record Dates: First submitted 2010-02-08; First posted 2010-07-26 (Estimated); Last update posted 2012-01-04 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer
Keywords: metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — genexol-PM; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Genexol-PM (Experimental): Genexol-PM 300mg/m2, diluted with 500ml of 5% dextrose or normal saline, intravenous infusion over 1 hour on day 1, every 3 week cycle.
  Interventions: Drug: Genexol-PM
- Paclitaxel (Active Comparator): Paclitaxel 175mg/m2, diluted with 500ml of 5% dextrose or normal saline, intravenous infusion over 3 hour on day 1, every 3 week cycle.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Genexol-PM — Treatment is given in the outpatient setting. Patients receive treatment every 3 weeks up to 6 cycles.
  Arms: Genexol-PM
Drug: Paclitaxel
  Arms: Paclitaxel

SUMMARY:
The purpose of this study is to evaluate the overall response rate of Genexol-PM compared with paclitaxel (cremophor-based paclitaxel) as palliative chemotherapy in anthracycline-pretreated patients with metastatic breast cancer.

DETAILED DESCRIPTION:
This is a prospective, two-armed, parallel group, randomized phase II study for the evaluation of Genexol-PM and paclitaxel. Up to 42 eligible patients will be enrolled in each treatment arm (a total of 84) according to the trial design. Patients will be randomly allocated to arm A (Genexol-PM) or arm B (Paclitaxel). They will be stratified by ER status(positive v negative), performance(ECOG 0 or 1 v 2), and prior adjuvant taxane (no v yes) The treatment will be continued up to 6 cycles, or will be discontinued before 6th cycle iin case of disease progression, unacceptable toxicity, or patient withdrawal. After discontinuation of study therapy, patients will proceed to the post-therapy follow-up phase of the study.

Patients may be enrolled in the study if they have documented measurable disease. Response will be documented by physical examination prior to each treatment cycle and a CT scan every two cycles or if disease progression is suspected. Responses will be assessed unidimensionally according to the RECIST. All partial or complete responses require confirmation with a second evaluation at least 4 weeks following the first documentation of response.

All toxicities encountered during the study will be evaluated before each cycle using the NCI CTC (National Cancer Institute Common Toxicity Criteria) version 3.0 scale. For peripheral neuropathy, the scale in Table 4 will be used to determine dose adjustments. Life-threatening toxicities should be reported immediately to the Study Chairman.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically diagnosed stage IV or recurrent breast cancer patients according to American Joint Committee on Cancer (AJCC 6th ed.)
2. Prior chemotherapy at least one anthracycline-containing regimen, in either adjuvant or metastatic setting is requested.
3. Previous hormonal therapy in adjuvant setting is allowed.
4. Previous adjuvant taxane chemotherapy in an adjuvant setting is allowed, if taxane-free interval is more than 12 months
5. previous chemotherapy for metastatic disease is not allowed except for the regimen including anthracycline.
6. Previous chemotherapy including taxane for metastatic disease is not allowed.
7. Prior radiation therapy is allowed as long as the irradiated area is not the only source of measurable disease.
8. No other forms of cancer therapy, such as radiation, immunotherapy or chemotherapy for at least 4 weeks before the enrollment in therapy.
9. Major surgery other than biopsy within the past two weeks.
10. At least 18 years old
11. Performance status of 0, 1 and 2 on the ECOG criteria.
12. Disease status must be that of measurable disease defined as RECIST:

    Lesions that can be accurately measured in at least one dimension > 10 mm with chest x-ray, spiral CT scan, MRI, or physical examination
13. Estimated life expectancy of at least 12 weeks.
14. Patient compliance that allow adequate follow-up.
15. Adequate major organ function including the following:

    ①Hematologic function: WBC ³ 3,000/mm3 or absolute neutrophil count (ANC) ³ 1,500/mm3, platelet count ³ 100,000/mm3

    ②Hepatic function: bilirubin 1.5 x UNL , AST/ALT levels 2.5 x UNL

    ③Renal function: serum creatinine 1.5mg/dL
16. Grade of baseline neuropathy should not be more than grade 1 by NCI CTC v.3.0
17. Patients should sign an informed consent
18. women of childbearing age should use non-hormonal contraceptive method.

Exclusion Criteria:

1. Serious concurrent infection or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complication of study therapy
2. Other malignancy with the past 5 years except adequately treated cutaneous basal cell carcinoma or uterine cervix in situ cancer
3. Psychiatric disorder that would preclude compliance.
4. uncontrolled CNS disease (eligible if the CNS disease is controlled with radiotherapy or corticosteroid)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-07; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
overall response rate | 21Aug2007~22Aug2008

CONTACTS AND LOCATIONS:
Overall Officials: Jungsil Ro, Ph,D, Principal Investigator — National Cancer Center, Korea